CLINICAL TRIAL: NCT00149084
Title: Pharmacogenomics-Based Tailor-Made Strategy for Eradication of Helicobacter Pylori
Brief Title: Tailored Treatment of H. Pylori Infection Based Polymorphisms of CYP2C19 and 23S rRNA of H. Pylori
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Collaborators: Yokoyama Foundation for Clinical Pharmacology (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Hp.CYP.001
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-09

CONDITIONS: Helicobacter Infections; Gastritis; Gastric Ulcer; Duodenal Ulcer
Keywords: The tailored H. pylori eradication therapy; CYP2C19 genotype; 23S rRNA; clarithromycin; Lansoprazole; Amoxicillin; H. pylori infection
MeSH Terms: conditions — Helicobacter Infections; Gastritis; Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole; Clarithromycin; Amoxicillin

INTERVENTIONS:
Drug: Lansoprazole, clarithromycin, amoxicillin

SUMMARY:
The eradication rate of the standard H. pylori eradication therapy (such as the triple therapy with a proton pump inhibitor [PPI], amoxicillin and clarithromycin) depends on bacterial susceptibility to clarithromycin and genotypes of CYP2C19 in patients. The investigators intend to investigate whether the tailored therapy based on the two above-mentioned factors increases the cure rate of the initial eradication therapy.

DETAILED DESCRIPTION:
Current treatment strategies for the eradication of H. pylori include a proton pump inhibitor (PPI) and one or two anti-bacterial agents, such as amoxicillin, clarithromycin, and metronidazole.

PPIs, such as lansoprazole and omeprazole, are mainly metabolized in the liver by a genetically determined enzyme, S-mephenytoin 4'-hydroxylase (CYP2C19). Plasma concentrations of PPIs and their activity for acid inhibition depend to a significant extent on the genetic differences in the activity of this enzyme. The acid inhibition attained by the standard dose of a PPI is sometimes therapeutically insufficient in individuals with the rapid extensive metabolizer (RM) genotype of CYP2C19, whereas that in individuals with poor metabolizer (PM) genotype of CYP2C19 is in most cases clinically sufficient. We have reported that the CYP2C19 genotype status is one of the determinants of H. pylori eradication therapy. In the triple therapy with a PPI, amoxicillin, and clarithromycin, bacterial susceptibility to clarithromycin as well as the CYP2C19 genotype status was significantly related to eradication rates of H. pylori. Therefore, the tailored treatment based on these two factors is expected to increase the eradication rates of the initial therapy.

Interestingly, both of CYP2C19 genotypes and bacterial susceptibility to clarithromycin can be measured by the genetic test of the single nucleotide polymorphisms (SNPs) of the CYP2C19 gene and the 23S rRNA gene of H. pylori, respectively. We have recently developed the inexpensive and reliable high-throughput method for measurement of such SNPs by the invader assay. Polymorphisms of CYP2C19 of patients and mutations of 23S rRNA of H. pylori associated with susceptibility to clarithromycin can be detected from the gastric tissue samples infected with H. pylori, such as the gastric tissue sample already used for rapid urease test (RUT).

Then, we treat H. pylori-positive patients by the tailored regimen based on genotypes of CYP2C19 of patients and 23S rRNA of H. pylori or the standard regimen and test the therapeutic efficacy of this pharmacogenomics-based tailored strategy in a prospective manner.

Patients were randomly assigned to the standard or tailored regimen group with the use of a computer-generated randomization list based on a blocked randomization method.

Patients assigned to the standard regimen group were treated with 30 mg of lansoprazole bid, 400 mg of clarithromycin bid, and 750 mg of amoxicillin bid for one week, which had been approved under the Japanese formulary regulation regardless of any pharmacogenomic backgrounds of H. pylori-infected peptic ulcer patients.

In the tailored regimen group, patients infected with a clarithromycin-sensitive strain of H. pylori are treated with triple therapy consisting of clarithromycin 200 mg tid, amoxicillin 500 mg tid and the individualized doses of lansoprazole dose (i.e., 30 mg tid in RMs, 15 mg tid in IMs, and 15 mg bid in PMs) for one week, while patients infected with a clarithromycin-resistant strain of H. pylori are treated with dual therapy consisting of amoxicillin 500 mg qid and the individualzed dose of lansoprazole (i.e., 30 mg qid in RMs, 15 mg qid in IMs, and 15 mg bid in PMs) for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H. pylori infection

Exclusion Criteria:

* Patients without H. pylori infection

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296
Dates: Start 2003-04

PRIMARY OUTCOMES:
Whether the tailored treatment yields a higher eradication rate in comparison with the standard treatment

SECONDARY OUTCOMES:
Cost-effectiveness of the tailored strategy

CONTACTS AND LOCATIONS:
Overall Officials: Takahisa Furuta, MD, PhD, Study Chair — Center for Clinical Research, Hamamatsu University School of Medicine
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan

REFERENCES:
- [Background] Furuta T, Shirai N, Sugimoto M, Nakamura A, Hishida A, Ishizaki T. Influence of CYP2C19 pharmacogenetic polymorphism on proton pump inhibitor-based therapies. Drug Metab Pharmacokinet. 2005 Jun;20(3):153-67. doi: 10.2133/dmpk.20.153. PMID 15988117
- [Background] Furuta T, Sagehashi Y, Shirai N, Sugimoto M, Nakamura A, Kodaira M, Kenmotsu K, Nagano M, Egashira T, Ueda K, Yoneyama M, Ohashi K, Ishizaki T, Hishida A. Influence of CYP2C19 polymorphism and Helicobacter pylori genotype determined from gastric tissue samples on response to triple therapy for H pylori infection. Clin Gastroenterol Hepatol. 2005 Jun;3(6):564-73. doi: 10.1016/s1542-3565(04)00779-7. PMID 15952098
- [Background] Furuta T, Shirai N, Sugimoto M, Ohashi K, Ishizaki T. Pharmacogenomics of proton pump inhibitors. Pharmacogenomics. 2004 Mar;5(2):181-202. doi: 10.1517/phgs.5.2.181.27483. PMID 15016609
- [Background] Sugimoto M, Furuta T, Shirai N, Kajimura M, Hishida A, Sakurai M, Ohashi K, Ishizaki T. Different dosage regimens of rabeprazole for nocturnal gastric acid inhibition in relation to cytochrome P450 2C19 genotype status. Clin Pharmacol Ther. 2004 Oct;76(4):290-301. doi: 10.1016/j.clpt.2004.06.008. PMID 15470328
- [Background] Furuta T, Shirai N, Xiao F, Takashita M, Sugimoto M, Kajimura M, Ohashi K, Ishizaki T. High-dose rabeprazole/amoxicillin therapy as the second-line regimen after failure to eradicate H. pylori by triple therapy with the usual doses of a proton pump inhibitor, clarithromycin and amoxicillin. Hepatogastroenterology. 2003 Nov-Dec;50(54):2274-8. PMID 14696516
- [Background] Furuta T, Shirai N, Ohashi K, Ishizaki T. Therapeutic impact of CYP2C19 pharmacogenetics on proton pump inhibitor-based eradication therapy for Helicobacter pylori. Methods Find Exp Clin Pharmacol. 2003 Mar;25(2):131-43. doi: 10.1358/mf.2003.25.2.723687. PMID 12731459
- [Background] Furuta T, Shirai N, Xiao F, Ohashi K, Ishizaki T. Effect of high-dose lansoprazole on intragastic pH in subjects who are homozygous extensive metabolizers of cytochrome P4502C19. Clin Pharmacol Ther. 2001 Nov;70(5):484-92. doi: 10.1067/mcp.2001.119721. PMID 11719736
- [Background] Furuta T, Shirai N, Takashima M, Xiao F, Hanai H, Nakagawa K, Sugimura H, Ohashi K, Ishizaki T. Effects of genotypic differences in CYP2C19 status on cure rates for Helicobacter pylori infection by dual therapy with rabeprazole plus amoxicillin. Pharmacogenetics. 2001 Jun;11(4):341-8. doi: 10.1097/00008571-200106000-00009. PMID 11434512
- [Background] Furuta T, Shirai N, Takashima M, Xiao F, Hanai H, Sugimura H, Ohashi K, Ishizaki T, Kaneko E. Effect of genotypic differences in CYP2C19 on cure rates for Helicobacter pylori infection by triple therapy with a proton pump inhibitor, amoxicillin, and clarithromycin. Clin Pharmacol Ther. 2001 Mar;69(3):158-68. doi: 10.1067/mcp.2001.113959. PMID 11240980
- [Background] Furuta T, Takashima M, Shirai N, Xiao F, Hanai H, Ohashi K, Ishizaki T. Cure of refractory duodenal ulcer and infection caused by Helicobacter pylori by high doses of omeprazole and amoxicillin in a homozygous CYP2C19 extensive metabolizer patient. Clin Pharmacol Ther. 2000 Jun;67(6):684-9. doi: 10.1067/mcp.2000.106826. PMID 10872651
- [Background] Furuta T, Ohashi K, Kosuge K, Zhao XJ, Takashima M, Kimura M, Nishimoto M, Hanai H, Kaneko E, Ishizaki T. CYP2C19 genotype status and effect of omeprazole on intragastric pH in humans. Clin Pharmacol Ther. 1999 May;65(5):552-61. doi: 10.1016/S0009-9236(99)70075-5. PMID 10340921
- [Background] Furuta T, Ohashi K, Kamata T, Takashima M, Kosuge K, Kawasaki T, Hanai H, Kubota T, Ishizaki T, Kaneko E. Effect of genetic differences in omeprazole metabolism on cure rates for Helicobacter pylori infection and peptic ulcer. Ann Intern Med. 1998 Dec 15;129(12):1027-30. doi: 10.7326/0003-4819-129-12-199812150-00006. PMID 9867757